CLINICAL TRIAL: NCT02822235
Title: Real-world Data of Moderate to Severe Inflammatory Bowel Disease in Brazil: a Non-interventional, Multicenter Study to Evaluate Disease Control, Treatment Patterns, Burden of Disease and Quality of Life (RISE BR)
Brief Title: Non-interventional Study of Moderate to Severe Inflammatory Bowel Disease in Brazil
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4008; U1111-1178-66445 (Registry Identifier: WHO)
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's Disease: Participants with diagnosis of moderate to severe Crohn's disease (CD) for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1. Participants with active IBD and CD at Day 1 were followed up for 12 months in prospective phase.
  Interventions: Other: No Intervention
- Ulcerative Colitis: Participants diagnosed with diagnosis of moderate to severe ulcerative colitis (UC) for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1. Participants with active IBD and UC at Day 1 were followed up for 12 months in prospective phase.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The purpose of this study is to gather information regarding the population with moderate to severe inflammatory bowel disease (IBD), the burden of the disease, and understand their treatment patterns, particularly on the use of available biologic therapies.

DETAILED DESCRIPTION:
This is a non-interventional study to determine the rate of control of disease activity in moderate to severe inflammatory bowel disease (IBD) participants, with two parts: cross-sectional evaluation (Day 1) with retrospective data collection and a prospective 12-month evaluation for patients with active IBD at cross-sectional evaluation (Day 1).

The study enrolled 407 patients. This multicenter trial was conducted in Brazil. Retrospective data of previous IBD treatments (drug, dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years will be collected. Prospective data was collected for a period of 12 months in participants with active disease. UC participants, with no or light disease activity at Day 1 did not continue to 12-month follow up. CD participants, with no or light disease activity at Day 1 but with colonoscopy or calprotectin levels (i.e, calprotectin >200 ug/g) in the previous year suggestive of inadequate control of activity progressed to 12-month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. 18 years or older (at the time of diagnosis of moderate to severe UC or CD).
3. Diagnosis of moderate to severe CD or UC for at least 6 months prior to Day 1 appointment according the clinical or endoscopic \ criteria.
4. Has provided the written informed consent. For the prospective period, eligible participants should present at least one of the following criteria that will only be applied at Day 1:
5. For CD participants:

   * Harvey Bradshaw Index (HBI) ≥8 or
   * Crohn's Disease Activity Index (CDAI) ≥220 or Considering that for CD participants, the disease activity may not be clearly documented only with clinical data, some objective criteria may be considered as entry criteria for the 12-month prospective period:
   * Colonoscopy in the previous year suggestive of inadequate control of activity or,
   * Calprotectin levels in the previous year suggestive of inadequate control of activity (i.e, calprotectin >200 µg/g).
6. For UC: partial Mayo Score ≥5.

Note: Participants with colostomy and prospective period: Although clinical scales defined above are impacted by colostomy these participants will not be excluded from the protocol to ensure the assessment of different clinical presentations of the IBD. In addition, participants with colostomy must follow the same criteria as above to be eligible to the prospective phase.

Exclusion Criteria:

1. Indeterminate or not classified colitis.
2. Current or previous participation in interventional clinical trial (within the last 3 years). In addition, for the 12-month prospective period, participants will be excluded if:
3. Presenting mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
4. Hospitalized participants at Day 1.
5. Current off label treatment with Vedolizumab.

Study Discontinuation Criteria It will be considered a premature termination the situation in which the participant discontinues the participation, i.e. they are withdrawn from the study before completing the 12 months of follow up period (365 days ± 14 days from Day 1), due to any of the reasons listed below:

1. Withdrawal of consent: participants who for any reason withdraw the free and informed consent;
2. Lost to follow-up (no return of the participant on the expected date of visit - drop-out from the protocol);
3. Death;
4. Study termination;
5. Any situation that places the participant within one of the exclusion criteria.

Note: Participants who are eligible for the prospective period, it means, with active disease at Day 1 but who during the 12 months period presents disease remission and/or no activity disease condition, are allowed to continue the participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with moderate to severe Crohn's Disease (CD) or Ulcerative Colitis (UC) were observed.
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abner Augusto Lobão Neto Clinical Science, Study Director — Takeda
Locations (13):
- Brazil (13):
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Juiz de Fora, Minas Gerais
  - Curitiba, Paraná
  - Teresina, Piauí
  - Porto Alegre, Rio Grande do Sul
  - Botucatu, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
  - Rio de Janeiro
  - São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at the 14 investigative sites in Brazil from 11 October 2016 to 19 Feb 2018.
Pre-assignment Details: Participants diagnosed with infectious bowel disease (IBD)- Crohn's disease (CD) or ulcerative colitis (UC) were observed to collect the retrospective data on Day 1. Participants with active disease at Day 1 entered Prospective phase and were followed up for a period of 12 months.
Groups:
- Crohn's Disease: Participants with diagnosis of CD for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1. Participants with active CD at Day 1 were followed up for 12 months in prospective phase.
- Ulcerative Colitis: Participants with diagnosis of UC for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1. Participants with active UC at Day 1 were followed up for 12 months in prospective phase.
Period: Cross-sectional Phase (Day 1)
Arm/Group | Crohn's Disease | Ulcerative Colitis
Started | 264 | 143
Completed (Participants with moderate to severe IBD at Day 1) | 118 | 36
Not Completed | 146 | 107
Not completed — Not Eligible for Prospective Follow-up | 144 | 107
Not completed — Reason Not Specified | 2 | 0
Period: Prospective Phase (Day 1 up to Month 12)
Arm/Group | Crohn's Disease | Ulcerative Colitis
Started | 118 | 36
Completed | 107 | 34
Not Completed | 11 | 2
Not completed — Withdrawal of Consent | 0 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Death | 1 | 0
Not completed — Reason Not Specified | 6 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who had completed the Day 1 assessment (occurred 6 months after start of enrolment), included in Cross-sectional population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crohn's Disease | Ulcerative Colitis | Total
Number analyzed (Participants) | 264 | 143 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (12.96) | 45.9 (13.83) | 43.9 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 81 | 224
  Male | 121 | 62 | 183
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 264 | 143 | 407
Professional Situation [Count of Participants; unit: Participants] — Participants were stratified by the following categories: employed, unemployed, student, retired, other, unknown.
  Participants
    Employed | 101 | 53 | 154
    Unemployed | 61 | 33 | 94
    Student | 10 | 5 | 15
    Retired | 30 | 15 | 45
    Other | 26 | 18 | 44
    Unknown | 36 | 19 | 55
Educational Level [Count of Participants; unit: Participants] — Participants were stratified by the following categories: not literate, primary school, primary school not completed, secondary school, secondary school not completed, higher education, higher education not completed, post-graduate/master of business administration (MBA), unknown.
  Participants
    Not Literate | 3 | 0 | 3
    Primary School | 26 | 11 | 37
    Primary School Not Completed | 26 | 27 | 53
    Secondary School | 74 | 33 | 107
    Secondary School Not Completed | 9 | 4 | 13
    Higher Education | 46 | 14 | 60
    Higher Education Not Completed | 18 | 8 | 26
    Post-graduate/Master of Business Administration | 5 | 1 | 6
    Unknown | 57 | 45 | 102
Income [Count of Participants; unit: Participants] — Participants were stratified by their monthly salary (MS). The following categories were made: >10-20 MS (R$ 8.800,01- R$ 17.600,00), >5-10 MS (R$ 4.400,01 - R$ 8.800,00), >3-5 MS (R$ 2.640,01 - R$ 4.440,00), >2-3 MS (R$ 1.760,01 - R$ 2.640,00), >1-2 MS (R$ 880,01 - R$ 1.760,00), >1/2-1 MS (R$ 440,01 - R$ 880,00), ≤1/2 MS (Until R$ 440,00 (including)), no income, unknown/not informed.
  Participants
    >10-20 MS (R$ 8.800,01- R$ 17.600,00) | 5 | 2 | 7
    > 5-10 MS (R$ 4.400,01 - R$ 8.800,00) | 8 | 7 | 15
    >3-5 MS (R$ 2.640,01 - R$ 4.440,00) | 28 | 10 | 38
    >2-3 MS (R$ 1.760,01 - R$ 2.640,00) | 25 | 12 | 37
    >1-2 MS (R$ 880,01 - R$ 1.760,00) | 49 | 16 | 65
    >1/2-1 MS (R$ 440,01 - R$ 880,00) | 18 | 7 | 25
    ≤1/2 MS (Until R$ 440,00 (Including)) | 1 | 1 | 2
    No Income | 25 | 14 | 39
    Unknown/Not Informed | 105 | 74 | 179
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with data available for height.
  cm
    number analyzed (Participants) | 250 | 136 | 386
    (all) | 166.0 (9.89) | 165.1 (10.70) | 165.7 (10.18)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with data available for weight.
  kg
    number analyzed (Participants) | 262 | 141 | 403
    (all) | 69.0 (14.52) | 70.1 (14.33) | 69.4 (14.45)
(Body Mass Index) BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index=weight (kg)/[height (m)^2] Population: Number analyzed is the number of participants with available for BMI.
  kg/m^2
    number analyzed (Participants) | 249 | 136 | 385
    (all) | 25.1 (4.67) | 25.7 (4.63) | 25.3 (4.66)
Smoking Status [Count of Participants; unit: Participants] — Participants were stratified by the following categories: never smoked, former smoker (not smoking at Day 1 but smoked 100 cigarettes in his/her lifetime), current smoker (smoking at Day 1 and has smoked 100 cigarettes in his/her lifetime), unknown.
  Participants
    Never Smoked | 171 | 91 | 262
    Former Smoker | 47 | 38 | 85
    Current Smoker | 24 | 3 | 27
    Unknown | 22 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Active Crohn's Disease (CD) at Day 1
Description: Participants with Harvey Bradshaw Index (HBI) score of ≥8 or Crohn´s Disease Activity Index (CDAI) ≥220 points at Day 1 were classified as participants with active disease. HBI scale assessed five dimensions (general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications). These dimensions were scored from the previous day. The total score ranges from 0 to 25. The CDAI evaluated the severity of signs and symptoms of CD. Collected data included information on the number of liquid stools, intensity of abdominal pain, general well-being, presence of comorbid conditions, use of medications for diarrhea, physical examination, and laboratory findings (abdominal mass, hematocrit, body weight), yielding 8 items that were combined with data from a 7-day diary to obtain the total CDAI score which ranges from 0 to approximately 600 points, where higher score indicates higher disease activity.
Time Frame: Day 1
Population: Cross-sectional population included all participants who had completed the Day 1 assessment (occurred 6 months after start of enrolment). Participants with CD from cross-sectional population were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 264
percentage of participants
  HBI Score ≥8: number analyzed (Participants) | 230
  HBI Score ≥8 | 16.52
  CDAI Score ≥220: number analyzed (Participants) | 77
  CDAI Score ≥220 | 25.97

2. Primary Outcome: Number of Participants With Active Ulcerative Colitis (UC) at Day 1
Description: Participants with ≥5 points in Partial Mayo Score were classified as active UC disease. The mayo score without endoscopy measured severity of ulcerative colitis. Three sub-scores for stool frequency, rectal bleeding, and physician's global assessment were each graded from 0 to 3 with higher scores indicating more severe disease. Individual sub-scores were then summed to provide the total score ranging from 0 (normal or inactive disease) to 9 (severe disease).
Time Frame: Day 1
Population: Cross-sectional population included all participants who had completed the Day 1 assessment (occurred 6 months after start of enrolment). Participants with UC from cross-sectional population were analyzed for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Ulcerative Colitis
Number analyzed (Participants) | 141
participants | 36

3. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Stratified by Age, Gender, Professional Status, Family History, Educational Level and Income at Day 1
Time Frame: Day 1
Population: Participants with moderate to severe CD or UC from the cross-sectional population, including all participants who had completed the Day 1 assessment (occurred 6 months after start of enrolment).
Measure: Count of Participants; unit: Participants
Groups:
- Crohn's Disease (Moderate to Severe Activity): Participants with diagnosis of moderate to severe Crohn's disease (CD) for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1. Participants with active CD at Day 1 were followed up for 12 months in prospective phase.
- Ulcerative Colitis (Moderate to Severe Activity): Participants with diagnosis of moderate to severe ulcerative colitis (UC) for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1. Participants with active UC at Day 1 were followed up for 12 months in prospective phase.
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
Participants
  Age ≥18-39 years old | 52 | 15
  Age ≥40-59 years old | 49 | 15
  Age ≥ 60 years old | 17 | 6
  Gender, Male | 49 | 10
  Gender, Female | 69 | 26
  Professional Status, Employed | 36 | 5
  Professional Status, Unemployed | 31 | 8
  Professional Status, Student | 2 | 3
  Professional Status, Retired | 13 | 6
  Professional Status, Other | 16 | 9
  Professional Status, Unknown | 20 | 5
  Family History of IBD | 15 | 2
  Educational Level, Not Literate | 1 | 0
  Educational Level, Primary School | 7 | 3
  Educational Level, Primary School Not Completed | 16 | 6
  Educational Level, Secondary School | 34 | 5
  Educational Level, Secondary School Not Completed | 3 | 2
  Educational Level, Higher Education | 23 | 2
  Educational Level, Higher Education Not Completed | 6 | 3
  Educational Level, Post-Graduate/MBA | 3 | 0
  Educational Level, Unknown | 25 | 15
  Income, >10-20 MS (R$ 8.800,01 - R$ 17.600,00) | 3 | 1
  Income, >5-10 MS (R$ 4.400,01 - R$ 8.800,00) | 1 | 1
  Income, >3-5 MS (R$ 2.640,01 - R$ 4.440,00) | 13 | 1
  Income, >2-3 MS (R$ 1.760,01 - R$ 2.640,00) | 10 | 1
  Income, >1-2 MS (R$ 880,01 - R$ 1.760,00) | 19 | 2
  Income, >½-1 MS (R$ 440,01 - R$ 880,00) | 10 | 2
  Income, ≤½ MS (Until R$ 440,00 (Including)) | 1 | 0
  Income, No Income | 10 | 6
  Income, Unknown | 31 | 10
  Income, Not Informed | 20 | 12

4. Secondary Outcome: Number of Participants With Moderate to Severe CD or UC Stratified by Clinical Variables
Description: Clinical variables included IBD type:CD/UC; anthropometric (Height, Weight and BMI); Family history; Smoking habits; Medical History/Comorbidities; Disease location -L1=ileal, L2=colonic disease, L3=ileocolic, L4=isolated upper GI tract disease location. Behavior as B1/B1+P=Non stenosing/non penetrating or B1+P=Non stenosing/non penetrating+perianal disease, B2/B2+P=Stenosing/B2+P=Stenosing+perianal disease B3/B3+P=Penetrating, B3+P=Penetrating+perianal disease, P=Penetrating disease. Extension of inflammation as E1=distal UC: proctitis or E1=distal UC: proctosigmoiditis extension of inflammation E2/E3=left-sided: mucosa inflammation extending up to splenic flexure or E3=pancolitis: mucosa inflammation up to proximal transverse colon and beyond extension of inflammation and severity of UC as S0=Clinical remission, S1=Mild UC, S2=Moderate UC, S3=Severe UC. Steroid behavior; Colonoscopy, Calprotectin levels >200ug/g, Eligibility for 12-month follow-up.
Time Frame: Day 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
Participants
  CD or UC, Moderate to Severe Activity | 118 | 36
  Height (cm) | NA — Data was not collected according to the pre-defined categories. | NA — Data was not collected according to the pre-defined categories.
  Weight (kg) | NA — Data was not collected according to the pre-defined categories. | NA — Data was not collected according to the pre-defined categories.
  BMI - <24 Kg/m^2: number analyzed (Participants) | 110 | 35
  BMI - <24 Kg/m^2 | 54 | 23
  BMI - 25 - 30 Kg/m^2: number analyzed (Participants) | 110 | 35
  BMI - 25 - 30 Kg/m^2 | 43 | 7
  BMI - ≥30 Kg/m^2: number analyzed (Participants) | 110 | 35
  BMI - ≥30 Kg/m^2 | 13 | 5
  Family History of IBD: number analyzed (Participants) | 94 | 32
  Family History of IBD | 15 | 2
  Smoking Status, Never Smoked: number analyzed (Participants) | 106 | 34
  Smoking Status, Never Smoked | 84 | 25
  Smoking Status, Former Smoker: number analyzed (Participants) | 106 | 34
  Smoking Status, Former Smoker | 15 | 9
  Smoking Status, Current smoker: number analyzed (Participants) | 106 | 34
  Smoking Status, Current smoker | 7 | 0
  Medical History, Comorbidity or EIM | 66 | 20
  Location of CD, L1: number analyzed (Participants) | 118 | 0
  Location of CD, L1 | 22 |
  Location of CD, L1+L4: number analyzed (Participants) | 118 | 0
  Location of CD, L1+L4 | 4 |
  Location of CD, L2: number analyzed (Participants) | 118 | 0
  Location of CD, L2 | 21 |
  Location of CD, L3: number analyzed (Participants) | 118 | 0
  Location of CD, L3 | 70 |
  Location of CD, L3+L4: number analyzed (Participants) | 118 | 0
  Location of CD, L3+L4 | 1 |
  Behavior, B1: number analyzed (Participants) | 118 | 0
  Behavior, B1 | 26 |
  Behavior, B1+P: number analyzed (Participants) | 118 | 0
  Behavior, B1+P | 5 |
  Behavior, B2: number analyzed (Participants) | 118 | 0
  Behavior, B2 | 39 |
  Behavior, B2+P: number analyzed (Participants) | 118 | 0
  Behavior, B2+P | 13 |
  Behavior, B3: number analyzed (Participants) | 118 | 0
  Behavior, B3 | 11 |
  Behavior, B3+P: number analyzed (Participants) | 118 | 0
  Behavior, B3+P | 24 |
  Extent Inflammation, E1-Distal: Proctitis: number analyzed (Participants) | 0 | 36
  Extent Inflammation, E1-Distal: Proctitis |  | 5
  Extent Inflammation, E1-Distal: Proctosigmoiditis: number analyzed (Participants) | 0 | 36
  Extent Inflammation, E1-Distal: Proctosigmoiditis |  | 5
  Extent of Inflammation, E2-Left-sided: number analyzed (Participants) | 0 | 36
  Extent of Inflammation, E2-Left-sided |  | 8
  Extent of Inflammation, E3-Pancolitis: number analyzed (Participants) | 0 | 36
  Extent of Inflammation, E3-Pancolitis |  | 18
  Severity, S1-Mild UC: number analyzed (Participants) | 0 | 36
  Severity, S1-Mild UC |  | 3
  Severity, S2-Moderate UC: number analyzed (Participants) | 0 | 36
  Severity, S2-Moderate UC |  | 25
  Severity, S3-Severe UC: number analyzed (Participants) | 0 | 36
  Severity, S3-Severe UC |  | 8
  Steroid Behavior, Steroid-dependent: number analyzed (Participants) | 22 | 13
  Steroid Behavior, Steroid-dependent | 17 | 10
  Steroid Behavior, Steroid-refractory Disease: number analyzed (Participants) | 5 | 13
  Steroid Behavior, Steroid-refractory Disease | 5 | 3
  Colonoscopy | 104 | 29
  Calprotectin >200ug/g | 13 | NA — Calprotectin levels was not applicable for UC participants as established in the protocol.

5. Secondary Outcome: Percentage of Participants With Moderate to Severe CD or UC Who Used Various Types of Therapies for IBD in Previous 3 Years
Description: Therapies for IBD included aminosalicylates, steroids, immunossupressors, biologics, antibiotics, surgeries and others. One participant could use more than one therapy.
Time Frame: Within the previous 3 years including Day 1
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
percentage of participants
  Salycyclic Derivates | 16.9 | 75.0
  Corticosteroids | 14.4 | 36.1
  Immunosuppresors | 67.8 | 47.2
  Biologic Therapy | 66.9 | 30.6
  Antibiotics | 9.3 | 13.9
  Surgeries | 27.1 | 2.8
  Others | 5.9 | 16.7

6. Secondary Outcome: Percentage of Participants With Moderate to Severe CD or UC Treated With Biologic Therapy Within 3 Previous Years
Description: IBD types included CD and UC. Biologic therapies included treatment with infliximab, adalimumab, vedolizumab, certolizumab, golimumab and ustekimumab. One participant could use more than one biologic therapy.
Time Frame: Within the previous 3 years including Day 1
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
percentage of participants
  Infliximab | 33.1 | 16.7
  Adalimumab | 30.5 | 11.1
  Vedolizumab | 2.5 | 5.6
  Certolizumab | 0.8 | 0.0
  Ustekimumab | 0.8 | 0.0

7. Secondary Outcome: Percentage of Participants With Moderate to Severe CD or UC Who Have Not Responded Previously to Biologic Therapies
Description: IBD types included CD and UC. Biologic therapies included treatment with infliximab, adalimumab, vedolizumab, certolizumab, golimumab and ustekimumab.
Time Frame: Day 1
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
percentage of participants | 36.4 | 33.3

8. Secondary Outcome: Percentage of Participants With Moderate to Severe CD or UC Who Were Ongoing IBD Treatment at Day 1
Description: Participants with moderate to severe CD or UC ongoing IBD treatment at Day 1 were reported.
Time Frame: Day 1
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
percentage of participants | 94.1 | 88.9

9. Secondary Outcome: Number of Participants With Moderate to Severe Activity of CD or With Light or no Activity Stratified by Socio-demographic Variables
Description: Socio-demographic variables included gender and professional status.
Time Frame: Day 1
Population: Cross-sectional population included all participants who had completed the Day 1 assessment (occurred 6 months after start of enrolment).
Measure: Count of Participants; unit: Participants
Groups:
- Crohn's Disease (Moderate to Severe Activity): Participants with diagnosis of moderate to severe Crohn's disease (CD) for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1. Participants with active IBD and CD at Day 1 were followed up for 12 months in prospective phase.
- Crohn's Disease (Mild or No Activity): Participants with diagnosis of mild Crohn's disease (CD) for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1.
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Crohn's Disease (Mild or No Activity)
Number analyzed (Participants) | 118 | 146
Participants
  Gender, Male | 49 | 72
  Gender, Female | 69 | 74
  Professional Status, Employed | 36 | 65
  Professional Status, Unemployed | 31 | 30
  Professional Status, Student | 2 | 8
  Professional Status, Retired | 13 | 17
  Professional Status, Other | 16 | 10
  Professional Status, Unknown | 20 | 16

10. Secondary Outcome: Number of Participants With Moderate to Severe Activity of CD or With Light or no Activity Stratified by Clinical Variables
Description: Clinical variables included IBD type:CD/UC; Family history; Smoking habits; Medical History/Comorbidities; Disease location -L1=ileal, L2=colonic disease, L3=ileocolic, L4=isolated upper GI tract disease location. Behavior as B1/B1+P=Non stenosing/non penetrating or B1+P=Non stenosing/non penetrating+perianal disease, B2/B2+P=Stenosing/B2+P=Stenosing+perianal disease B3/B3+P=Penetrating, B3+P=Penetrating+perianal disease, P=Penetrating disease. Steroid behavior; Colonoscopy, Calprotectin levels >200ug/g.
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Crohn's Disease (Mild or No Activity)
Number analyzed (Participants) | 118 | 146
Participants
  Family History of IBD | 15 | 18
  Smoking Status, Never Smoked: number analyzed (Participants) | 106 | 136
  Smoking Status, Never Smoked | 84 | 87
  Smoking Status, Former Smoker: number analyzed (Participants) | 106 | 136
  Smoking Status, Former Smoker | 15 | 32
  Smoking Status, Current smoker: number analyzed (Participants) | 106 | 136
  Smoking Status, Current smoker | 7 | 17
  Medical History, Comorbidity or EIM | 66 | 77
  Location of CD, L1: number analyzed (Participants) | 118 | 141
  Location of CD, L1 | 22 | 39
  Location of CD, L1+L4: number analyzed (Participants) | 118 | 141
  Location of CD, L1+L4 | 4 | 2
  Location of CD, L2: number analyzed (Participants) | 118 | 141
  Location of CD, L2 | 21 | 21
  Location of CD, L3: number analyzed (Participants) | 118 | 141
  Location of CD, L3 | 70 | 74
  Location of CD, L3+L4: number analyzed (Participants) | 118 | 141
  Location of CD, L3+L4 | 1 | 5
  Behavior, B1 | 26 | 20
  Behavior, B1+P | 5 | 7
  Behavior, B2 | 39 | 40
  Behavior, B2+P | 13 | 18
  Behavior, B3 | 11 | 23
  Behavior, B3+P | 24 | 33
  Behavior, P | 0 | 5
  Steroid Behavior, Steroid-dependent: number analyzed (Participants) | 22 | 25
  Steroid Behavior, Steroid-dependent | 17 | 14
  Steroid Behavior, Steroid-refractory disease: number analyzed (Participants) | 22 | 25
  Steroid Behavior, Steroid-refractory disease | 5 | 11
  Colonoscopy | 104 | 107
  Calprotectin >200ug/g | 41 | 38

11. Secondary Outcome: Percentage of Participants With Treatment Beginning or Ongoing at Day 1 by Moderate to Severe Activity of CD or With Light or no Activity Stratified by Treatment Variables
Description: Treatment variables included previous treatments or regimens (aminosalicylates, steroids, immunossupressors, biologics, antibiotics); and previous surgeries for IBD. One participant could use more than one treatment regimens.
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Crohn's Disease (Mild or No Activity)
Number analyzed (Participants) | 118 | 146
Participants
  Type of Therapy, Salicylic Derivates | 20 | 19
  Type of Therapy, Corticosteroids | 17 | 13
  Type of Therapy, Immunosuppressors | 80 | 98
  Type of Therapy, Biologic Therapy | 79 | 110
  Type of Therapy, Antibiotics | 11 | 3
  Type of Therapy, Other | 7 | 6
  Previous Surgery | 32 | 35

12. Secondary Outcome: Number of Participants With Moderate to Severe Activity of UC or With Light or no Activity Stratified by Socio-demographic Variables
Description: Socio-demographic variables included gender and professional status.
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- Ulcerative Colitis (Mild or No Activity): Participants with diagnosis of mild ulcerative colitis (UC) for at least 6 months prior to Day 1 were observed to collect the retrospective data including previous inflammatory bowel disease (IBD) treatments (drug dose, treatment duration, drug changes), and use of other health resources related with the management of IBD for previous three years at Day 1.
Arm/Group | Ulcerative Colitis (Moderate to Severe Activity) | Ulcerative Colitis (Mild or No Activity)
Number analyzed (Participants) | 36 | 107
Participants
  Gender, Male | 10 | 52
  Gender, Female | 26 | 55
  Professional Status, Employed | 5 | 48
  Professional Status, Unemployed | 8 | 25
  Professional Status, Student | 3 | 2
  Professional Status, Retired | 6 | 9
  Professional Status, Other | 9 | 9
  Professional Status, Unknown | 5 | 14

13. Secondary Outcome: Number of Participants With Moderate to Severe Activity of UC or With Light or no Activity Stratified by Clinical Variables
Description: Clinical variables included IBD type:CD/UC; Family history; Smoking habits; Medical History/Comorbidities; Extension of inflammation as E1=distal UC: proctitis or E1=distal UC: proctosigmoiditis extension of inflammation E2/E3=left-sided: mucosa inflammation extending up to splenic flexure or E3=pancolitis: mucosa inflammation up to proximal transverse colon and beyond extension of inflammation and severity of UC as S0=Clinical remission, S1=Mild UC, S2=Moderate UC, S3=Severe UC. Steroid behavior; Colonoscopy, Calprotectin levels >200ug/g.
Time Frame: Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Ulcerative Colitis (Moderate to Severe Activity) | Ulcerative Colitis (Mild or No Activity)
Number analyzed (Participants) | 36 | 107
Participants
  Family History of IBD | 2 | 13
  Smoking Status, Never Smoked: number analyzed (Participants) | 34 | 98
  Smoking Status, Never Smoked | 25 | 66
  Smoking Status, Former Smoker: number analyzed (Participants) | 34 | 98
  Smoking Status, Former Smoker | 9 | 29
  Smoking status, Current smoker: number analyzed (Participants) | 34 | 98
  Smoking status, Current smoker | 0 | 3
  Medical History, Comorbidity or EIM | 20 | 59
  Extent Inflammation, E1-Distal: Proctitis | 5 | 12
  Extent Inflammation, E1-Distal: Proctosigmoiditis | 5 | 21
  Extent of Inflammation, E2-Left-sided | 8 | 18
  Extent of Inflammation, E3-Pancolitis | 18 | 56
  Severity, S0-Clinical Remission | 0 | 57
  Severity, S1-Mild UC | 3 | 29
  Severity, S2-Moderate UC | 25 | 15
  Severity, S3-Severe UC | 8 | 6
  Steroid Behavior, Steroid-dependent: number analyzed (Participants) | 13 | 21
  Steroid Behavior, Steroid-dependent | 10 | 13
  Steroid Behavior, Steroid-refractory disease: number analyzed (Participants) | 13 | 21
  Steroid Behavior, Steroid-refractory disease | 3 | 8
  Colonoscopy | 29 | 87

14. Secondary Outcome: Percentage of Participants With Treatment Beginning or Ongoing at Day 1 by Moderate to Severe Activity of UC or With Light or no Activity Stratified by Treatment Variables
Description: Treatment variables include previous treatments or regimens (aminosalicylates, steroids, immunomodulators, immunossupressors, biologics, antibiotics); and previous surgeries for IBD. One participant could use more than one treatment regimens.
Time Frame: Day 1
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Ulcerative Colitis (Moderate to Severe Activity) | Ulcerative Colitis (Mild or No Activity)
Number analyzed (Participants) | 36 | 107
percentage of participants
  Type of Therapy, Salicylic Derivates | 75.0 | 68.2
  Type of Therapy, Corticosteroids | 36.1 | 12.1
  Type of Therapy, Immunosuppressors | 47.2 | 43.0
  Type of Therapy, Biologic Therapy | 30.6 | 28.0
  Type of Therapy, Antibiotics | 13.9 | 1.9
  Type of Therapy, Other | 16.7 | 7.9
  Previous Surgery | 2.8 | 2.8

15. Secondary Outcome: Harvey Bradshaw Index (HBI) Total Score in Participants Who Had Moderate to Severe Active CD at Day 1 and Month 12
Description: HBI scale assessed the severity of CD. HBI scale assessed five dimensions (general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications). These dimensions were scored from the previous day. The total score ranges from 0 to 25. Higher score indicates higher disease activity.
Time Frame: Day 1 and Month 12
Population: Longitudinal population included all participants who were eligible for the prospective period. Participants with active CD with data available for analysis at Day 1 and Month 12 were observed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 40
score on a scale
  Day 1: number analyzed (Participants) | 36
  Day 1 | 7.2 (8.53)
  Month 12 | 3.7 (3.68)

16. Secondary Outcome: Crohn´s Disease Activity Index (CDAI) Total Score in Participants Who Had Moderate to Severe Active CD at Day 1 and Month 12
Description: CDAI evaluated the severity of signs and symptoms of CD. Collected data included information on the number of liquid stools, intensity of abdominal pain, general well-being, presence of comorbid conditions, use of medications for diarrhea, physical examination, and laboratory findings (abdominal mass, hematocrit, body weight), yielding 8 items that were combined with data from a 7-day diary to obtain the total CDAI score which ranges from 0 to approximately 600 points, where higher score indicates higher disease activity.
Time Frame: Day 1 and Month 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 40
score on a scale
  Day 1: number analyzed (Participants) | 19
  Day 1 | 197.3 (124.44)
  Month 12: number analyzed (Participants) | 18
  Month 12 | 122.0 (68.82)

17. Secondary Outcome: Partial Mayo Score in Participants Who Had Moderate to Severe Active UC at Day 1 and Month 12
Description: The mayo score without endoscopy measured severity of ulcerative colitis. Three sub-scores for stool frequency, rectal bleeding, and physician's global assessment were each graded from 0 to 3 with higher scores indicating more severe disease. Individual sub-scores were then summed to provide the total score ranging from 0 (normal or inactive disease) to 9 (severe disease).
Time Frame: Day 1 and Month 12
Population: Longitudinal population included all participants who were eligible for the prospective period. Participants with active UC with data available for analysis at Day 1 and Month 12 were observed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 10
score on a scale
  Day 1 | 5.4 (0.52)
  Month 12 | 2.3 (2.16)

18. Secondary Outcome: Percentage of Participants With Moderate to Severe Active CD or UC Who Changed IBD Treatment at Month 12, by Reason
Description: One participant could have more than one reason for discontinuation.
Time Frame: Month 12
Population: Longitudinal population included all participants who were eligible for the prospective period (participants with active IBD at Day 1).
Measure: Number; unit: percentage of participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 111 | 36
percentage of participants
  Adverse Reaction | 7.1 | 3.8
  Comorbidity | 0.4 | 0.0
  Contraindication | 0.0 | 1.3
  Pregnancy | 0.4 | 3.2
  Surgery | 0.7 | 0.0
  Weight change | 0.4 | 0.0
  Poor Effectiveness | 10.6 | 12.4
  Remission | 11.0 | 27.5
  Patient decision | 1.8 | 5.0
  Patient poor adherence | 3.2 | 1.3
  Patient access to the treatment | 0.7 | 0.0
  Other | 25.1 | 2.5
  Unknown | 38.9 | 46.3

19. Secondary Outcome: Quality of Life as Assessed by European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Day 1
Description: EQ-5D questionnaire is an instrument used to measure general HRQOL in participants with IBD. Each dimension has three possible levels: 1 = none, 2 = moderate or 3 = extreme. The EQ-5D VAS score is a self-assigned rating of overall health using a 20-cm visual, vertical scale, with a score of 0 as the worst and 100 as the best possible health. An increase of ≥7 points in the EQ-5D VAS score represents a clinically meaningful improvement in quality of life for participants.
Time Frame: Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
score on a scale | 68.9 (22.14) | 55.2 (22.44)

20. Secondary Outcome: Quality of Life as Assessed by 36-Item Short Form Health Survey (SF-36) Component Score at Day 1
Description: The Short Form-36 (SF-36) is a questionnaire that evaluates a participant's health related quality of life. SF-36 includes 36 questions related to 8 health dimensions: physical functioning, role-physical (role limitations due to physical health problems), bodily pain, general health, vitality (energy/fatigue), social functioning, role-emotional (role limitations due to emotional problems), and mental health. Based on these 4 scales (physical functioning, role-physical, bodily pain, general health), the physical component summary (PCS) score is generated which ranges between 0 and 100, with higher scores indicating a better quality of life. Based on these 4 scales (vitality, social functioning, role-emotional, and mental health), the mental component summary (MCS) score is generated which ranges between 0 and 100, with higher scores indicating a better quality of life.
Time Frame: Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
score on a scale
  Mental Component Score | 42.6 (12.00) | 36.4 (13.48)
  Physical Component Score | 43.3 (10.15) | 40.8 (9.13)

21. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Day 1
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) was a 32-item questionnaire that measures 4 dimensions: bowel function, emotional status, systemic symptoms, and social function. Within dimensions, each question presented seven possible answers/points. Each domain score was the sum of 8 responses each ranging from 1 to 7, where 1 indicated worst function and 7 the best. The total score ranged from 32 to 224, with higher scores representing better quality of life. The IBDQ was not validated for participants with colostomies and therefore was not be applied for these participants.
Time Frame: Day 1
Population: Cross-sectional population included all participants who had completed the Day 1 assessment (occurred 6 months after start of enrolment). Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 263 | 142
score on a scale | 158.9 (41.41) | 153.2 (49.66)

22. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Domain Score at Day 1
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) was a 32-item questionnaire that measures 4 dimensions: bowel function, emotional status, systemic symptoms, and social function. Within dimensions, each question presented seven possible answers/points. Each domain score was the average of 8 responses each ranging from 1 to 7, where 1 indicated worst function and 7 the best function. The IBDQ was not validated for participants with colostomies and therefore was not be applied for these participants.
Time Frame: Day 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 263 | 142
score on a scale
  Bowel Systems | 5.4 (1.24) | 5.1 (1.63)
  Emotional Health | 4.7 (1.46) | 4.6 (1.64)
  Systemic Systems | 4.6 (1.48) | 4.5 (1.64)
  Social Function | 5.2 (1.58) | 5.0 (1.81)

23. Secondary Outcome: Mean of Percentage of Total Work Impairment Due to CD as Assessed by Work Productivity and Activity Impairment (WPAI) Questionnaire at Day 1
Description: The Work Productivity and Activity Impairment questionnaire (WPAI) assessed the impact of IBD on work productivity and daily activities during the previous 7 days. The 'impairment while working due to IBD' was calculated based on one question: to what degree did the disease impair the productivity while working in the past seven days from visit and the 'activity impairment' was calculated based on Question: how much did the disease affect ability to perform regular daily activities, other than work at a job? Percentage of overall work impairment due to IBD is calculated as: Absenteeism+(1-Absenteeism)*Presenteeism. The total score ranges from 0 (no impairment) to 100% (total loss of work productivity).
Time Frame: Day 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage of total work impairment
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 264 | 143
percentage of total work impairment
  Percentage of Total Work Productivity Impairment: number analyzed (Participants) | 97 | 50
  Percentage of Total Work Productivity Impairment | 32.3 (32.97) | 25.3 (33.13)
  Percentage of Total Activity Impairment: number analyzed (Participants) | 264 | 142
  Percentage of Total Activity Impairment | 35.8 (33.49) | 39.9 (37.45)

24. Secondary Outcome: Mean of Percentage of Work Time Missed Due to CD as Assessed by WPAI at Day 1
Description: Mean total activity impairment due to IBD from WPAI questionnaire was reported. The 'overall work impairment due to IBD' was calculated based on three items: (Q2) the number of hours missed from work due to health problems in the past seven days; (Q4) the number of actual work hours in the past seven days; and (Q5) to what degree did the disease impair the productivity while working past seven days. The data was calculated using the formula Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)] and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 98 | 50
percentage of work time missed | 12.6 (23.78) | 11.7 (26.69)

25. Secondary Outcome: Mean of Percentage of Impairment While Working Due to CD as Assessed by WPAI at Day 1
Description: Mean impairment while working due to IBD from WPAI questionnaire was reported. The 'impairment while working due to IBD' was calculated based on one item: (Q5) to what degree did the disease impair the productivity while working in the past seven days. The item was measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/ working). The data was calculated using the formula Q5/10 and converted to percent. ata are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 110 | 57
percentage of impairment while working | 24.4 (27.94) | 17.5 (26.00)

26. Secondary Outcome: Mean of Percentage of Total Activity Impairment Due to CD as Assessed by WPAI
Description: as for outcome 24
Time Frame: Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of total activity impairment
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 264 | 142
percentage of total activity impairment | 35.8 (33.49) | 39.9 (37.45)

27. Secondary Outcome: Percentage of Participants Who Used Healthcare Resources
Description: Healthcare resources used in the previous 3 years included imaging and laboratory testing, surgeries, hospitalizations, and consultations.
Time Frame: Day 1
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Crohn's Disease (Moderate to Severe Activity) | Ulcerative Colitis (Moderate to Severe Activity)
Number analyzed (Participants) | 118 | 36
percentage of participants
  Previous Imaging and Laboratory Testing Due to IBD | 98.3 | 100.0
  Previous Surgery for IBD | 27.1 | 2.8
  Previous Hospitalization Due to IBD | 43.2 | 30.6
  Previous Medical Appointments Due to IBD | 99.2 | 100.0

ADVERSE EVENTS:
Time Frame: Up to Month 12
Description: Data of adverse events or adverse drug reactions were not collected as part of the study database.
Arm/Group | Crohn's Disease | Ulcerative Colitis
All-Cause Mortality (participants affected / at risk) | 1/264 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Missing data on paticipants medical records in retrospective analysis and missing information in medical activity scores of participants in prospective analysis resulted in improper collection of data for IBD participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT02822235/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT02822235/SAP_001.pdf